CLINICAL TRIAL: NCT04098445
Title: TRANSPIRE: Lung Injury in a Longitudinal Cohort of Pediatric HSCT Patients
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0001C
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic Stem Cell Transplant (HSCT); Diffuse Alveolar Hemorrhage; Thrombotic Microangiopathies; Interstitial Pneumonitis; Bronchiolitis Obliterans
MeSH Terms: conditions — Thrombotic Microangiopathies; Lung Diseases, Interstitial; Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric and young adult HSCT recipients: Prospective multi-institutional cohort study in pediatric patients undergoing allogeneic (alloHSCT) or autologous hematopoietic stem cell transplantation (autoHSCT).

SUMMARY:
Hematopoietic stem cell transplant (HSCT) is an effective but toxic therapy and pulmonary morbidity affects as many as 25% of children receiving transplant. Early pulmonary injury includes diffuse alveolar hemorrhage (DAH), thrombotic microangiopathy (TMA) interstitial pneumonitis (IPS) and infection, while later, bronchiolitis obliterans is a complication of chronic GVHD associated with severe morbidity and mortality. Improved diagnosis and treatment of pulmonary complications are urgently needed as survival after HSCT improves, and as HSCT is increasingly used for non-malignant disorders such as sickle cell disease. Currently, there are large and important gaps in the investigator's knowledge regarding incidence, etiology and optimal treatment of pulmonary complications. Moreover, young children unable to perform spirometry are often diagnosed late, and strategies for monitoring therapeutic response are limited.

This is a prospective multi-institutional cohort study in pediatric patients undergoing allogeneic hematopoietic stem cell transplantation (alloHSCT). Assembly of a large prospective uniformly screened cohort of children receiving HSCT, together with collection of biological samples, will be an effective strategy to identify mechanisms of lung injury, test novel diagnostic strategies for earlier diagnosis, and novel treatments to reduce morbidity and mortality from lung injury after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≤ 24 years of age undergoing allogeneic or autologous HSCT.

Exclusion Criteria:

* Subjects over 24 years of age.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study participants will include eligible patients undergoing allogeneic or autologous HSCT at participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Lung Injury after HSCT | 24 months after HSCT
  Participants will be assessed for lung injury at 24 months after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (9):
- United States (9):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Dana-Farber Cancer Institute/Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Texas Children'S Hospital, Houston, Texas
  - Seattle Children'S Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Koo J, Cooper R, Edwards SL, Lane A, Loveless SK, Strecker L, Lake KE, Myers KC, Towe C, Patti J, Walkup LL, Wikenheiser-Brokamp KA, MacMillan ML, Lacher P, Griffin T, Tekman M, Cisneros GS, Wu K, Zinter MS, Urrego FA, Baker KS, Abts MF, Ballard S, Freedman JL, Caraballo A, Young LR, Josephson MB, Allen JL, Camburn DM, Doherty EE, Azamian MS, Arredondo M, Silva-Carmona M, Lehmann LE, Wong W, Gaffin JM, McAlpine W, Li M, Goldfarb SB, Woods JC, Davies SM. High Prevalence of Abnormal Baseline Lung Function in Pediatric and Young Adult Hematopoietic Stem Cell Transplant Recipients: A Report from the TRANSPIRE Study. Pediatr Blood Cancer. 2025 Oct;72(10):e31916. doi: 10.1002/pbc.31916. Epub 2025 Jul 21. PMID 40692216